CLINICAL TRIAL: NCT00641511
Title: Pharmacogenetic Clinical Trial of Nepicastat for PTSD
Brief Title: Pharmacogenetic Clinical Trial of Nepicastat for Post Traumatic Stress Disorder (PTSD)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Houston site withdrew as a study site.
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Tuscaloosa Veterans Affairs Medical Center (U.S. Federal Agency); Ralph H. Johnson VA Medical Center (U.S. Federal Agency); Acorda Therapeutics (Industry)
Responsible Party: Principal Investigator, Thomas Kosten, MD, , Waggoner Chair and Professor of Psychiatry, Neuroscience, Pharmacology, Immunology & Pathology, Michael E. DeBakey VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H22601; Inv117-Kosten-CL01
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Post Traumatic Stress Disorder (PTSD)
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — nepicastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Medication arm - SYN117 aka Nepicastat) (Experimental): Veterans will be receiving the study medication Nepicastat initiated with a 3-day loading phase of 40 mg on day 1, 80 mg on day 2 and 120 mg on day 3 (orally) and be continued at 120 mg once daily; During the 8 weeks (weeks: 7-14) extension phase, those from both treatment groups of the RCT phase will start open-label, active Nepicastat (i.e. no chance of placebo) treatment and be followed for an additional 8 weeks. Those who have a prior defined positive clinical response to the study medication, Nepicastat, will be continued on open label Nepicastat at 120mg once daily, in order to assess further improvement and safety; those who do not have a positive clinical response during the 6 weeks RCT will be offered the addition of the standard first-line PTSD pharmacotherapy, Paroxetine. Paroxetine is an allowed concomitant medication (i.e. "rescue medication") and is not considered a research medication or subject of a research question during the 8 weeks extension phase.
  Interventions: Drug: SYN117 (nepicastat)
- 2 (Placebo arm) (Placebo Comparator): During the 6 weeks ( weeks: 1-6) double- blind, randomized clinical trial (RCT) phase, the veterans who have been randomized to the placebo treatment group will be receiving placebo pills. During the 8 weeks (weeks: 7-14) extension phase, all veterans from both treatment groups of the RCT phase will start open-label, active Nepicastat (i.e. no chance of placebo) treatment and be followed by the study team for an additional 8 weeks. The veterans on the placebo during the RCT will receive the study medication at end of the study week 6, the medication will be initiated with a 3-day loading phase of 40 mg on day 1, 80 mg on day 2 and 120 mg on day 3 (orally) and be continued at 120 mg once daily for 8 weeks until the end of the study.
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: SYN117 (nepicastat) — 120 mg per day
  Other Names: nepicastat
  Arms: 1 (Medication arm - SYN117 aka Nepicastat)
Drug: Placebo comparator — once per day placebo capsules
  Arms: 2 (Placebo arm)

SUMMARY:
Assess the effect of nepicastat in the treatment of in Post Traumatic Stress Disorder (PTSD) in conflict or combat zone experienced veterans, in comparison to placebo.

DETAILED DESCRIPTION:
The primary treatment objective is to assess the global efficacy of nepicastat in the treatment of hyper-arousal in Post Traumatic Stress Disorder (PTSD) in conflict or combat zone experienced veterans, in comparison to placebo. The secondary treatment objectives are to assess the ability of nepicastat to induce PTSD remission; treat PTSD and other PTSD symptom clusters and improve quality of life and overall functioning. A medical safety objective is to assess the tolerability and side effects of nepicastat in the treatment of PTSD in veterans who served in conflict zones at least one time between 1990 -2008 [includes Operation Iraqi Freedom/Operation Enduring Freedom (OIF/OEF), Afghanistan, Gulf War, etc .

This is a 6-week study with the long-term objective is to define the best approach to treating PTSD and enhancing the quality of life in patients. Results from this pilot study will assist clinicians in treating active military service members or veterans with PTSD by developing new treatment algorithms for future larger studies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Patient understands the risks and benefits and agrees to visit frequency and procedures
3. Male or female
4. Any race or ethnic origin
5. Served in conflict zones at least one time between 1990 -2008 [includes Operation Iraqi Freedom/Operation Enduring Freedom (OIF/OEF), Afghanistan, Gulf War, etc]
6. Currently Active Duty, National Guard, Reservist, Veteran, and/or Retired Military
7. DSM-IV Diagnosis of Post-Traumatic Stress Disorder (PTSD)
8. No substance use disorders (except for nicotine and caffeine) in the previous 2 months
9. Free of psychotropic medication for 2 weeks prior to randomization (a low dose sedative hypnotic is allowed for severe insomnia if used sparingly)
10. Physical and laboratory panel are within normal limits or not clinically significant
11. Women of childbearing potential must be using medically-approved methods of birth control
12. 18 to 65 years of age

Exclusion Criteria:

1. Lifetime history of bipolar I, schizophrenia, schizoaffective or cognitive disorders
2. Actively considering plans of suicide or homicide
3. Psychotic symptoms that in the investigator's opinion impair the patient's ability to give informed consent or make it unsafe for patient to be maintained without a neuroleptic
4. Unstable general medical conditions or a contraindication to the use of nepicastat
5. Intolerable side effects or allergic reaction to nepicastat
6. Women planning to become pregnant or breastfeed during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in CAPS(D) hyperarousal scores as compared to placebo | 6 weeks

SECONDARY OUTCOMES:
Change from baseline in Structured Interview of Posttraumatic Stress Disorder (SIP) as compared to placebo | 6 weeeks
Change from baseline in Montgomery Asberg Depression Rating Scale (MADRS)as compared to placebo | 6 weeks
Clinicians global impression of Severity and Improvement | 6 weeks
Quality of life assessment as measured by the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q). | 6 weeks
Change from baseline in Davidson Trauma Scale (DTS) as compared to placebo | 6 weeks
Change from baseline in Sheehan Disability Scale as compared to placebo | 6 weeks
Change from baseline in Clinician Administered PTSD Scale- Symptom (CAPS-SX) as compared to placebo | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kosten, MD, Study Chair — Baylor College of Medicine, and DeBakey VAMC; Lori Davis, MD, Study Director — Tuscaloosa VAMC; Mark Hamner, MD, Principal Investigator — Ralph H Johnson VAMC; David P. Graham, MD, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (3):
- United States (3):
  - Tuscaloosa VAMC, Tuscaloosa, Alabama
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Michael E. Debakey VAMC, Houston, Texas